CLINICAL TRIAL: NCT01862484
Title: Neuroimaging of Diet and Medication in the Treatment of ADHD
Brief Title: Neuroimaging of Diet in ADHD: Phase I
Acronym: FTF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Steven Pliszka, Professor and Chief, Division of Child and Adolescent Psychiatry, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21MH09680
Record Dates: First submitted 2013-05-17; First posted 2013-05-24 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Diet; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restricted Diet (Experimental): Child is on an additive, gluten free diet. Child receives daily snacks which conform to the restrictive diet.
  Interventions: Dietary Supplement: Restricted Diet
- Ruse Diet (Sham Comparator): Child is on an additive, gluten free diet. Child receives daily snacks which violate the restrictive diet.
  Interventions: Dietary Supplement: Ruse Diet

INTERVENTIONS:
Dietary Supplement: Restricted Diet — Child is on an additive, gluten free diet. Child receives daily snacks which conform to the restrictive diet.
  Arms: Restricted Diet
Dietary Supplement: Ruse Diet — Child is on an additive, gluten free diet. Child receives daily snacks which violate the restrictive diet
  Arms: Ruse Diet

SUMMARY:
Children with Attention Deficit Hyperactivity Disorder (ADHD) aged 9-12 years of age will be placed on a restriction diet for a 5 week period. Children will be randomized to either receive daily snacks that conform to the diet or will violate the diet (Ruse diet) in a double blind fashion. It is hypothesized that children who are consistently on the restricted diet (relative to those on the ruse diet) will show improvements in ADHD symptoms.

DETAILED DESCRIPTION:
The ADHD rating scale (RS) will be the principal behavioral outcome measure. We hypothesize that children on restriction diet will have significantly lower ADHD RS scores after 5 weeks relative to the Ruse diet group. In addition children will undergo functional magnetic resonance imaging (fMRI) at baseline and again at 5 weeks. Children will perform a flanker task known to engage the dorsolateral prefrontal cortex (DLPFC) and the anterior cingulate cortex (ACC) during attention tasks. The children will also perform will look at pictures of appealing and unappealing food and rate whether they would like to eat it or not. This task is known to activate the ventral striatum (VS) (reward processing). A secondary hypothesis is whether children on the restricted diet will show changes in activity and connectivity of areas (DLPFC, ACC, VS) relative to those on the Ruse diet.

ELIGIBILITY:
Inclusion Criteria:

* Age 9-12 years
* Meets criteria for Attention Deficit Hyperactivity Disorder
* Parent must agree to use Study Diet Manual

Exclusion Criteria:

* Any Axis I psychiatric disorder other than Oppositional Defiant Disorder or Anxiety Disorder not requiring psychopharmacological management
* Not currently on any pharmacological agent other than medication for ADHD

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stevn R Pliszka, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited through advertisement in magazines and flyers posted in child psychiatry clinics
Pre-assignment Details: 40 children were enrolled, a total of 29 were randomized. Of the remaining 11, 8 were screen failures, 3 withdrew from the study prior to randomization.
Period: Overall Study
Arm/Group | Restricted Diet | Ruse Diet
Started | 15 | 14
Completed | 13 | 6
Not Completed | 2 | 8
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Population: Children age 9 to 12 with ADHD.
Groups:
- Total: Total of all reporting groups
Arm/Group | Restricted Diet | Ruse Diet | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 14 | 29
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (1.73) | 10.83 (1.25) | 10.82 (1.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 9 | 10
  Male | 14 | 5 | 19
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: ADHD Rating Scale IV
Description: The ADHD Rating Scale is an 18 items scale containing items related to the diagnosis of Attention Deficit Hyperactivity Disorder (ADHD). It is filled out by the parent. Each item is rated 0-3, the range of scores is 0 to 54, with 25 being the score below which the patient is considered to be in remission. Reference: DuPaul GJ, Power TJ, Anastopoulos AD, Reid R: ADHD Rating Scales-IV: Checklists, Norms and Clinical Interpretation. New York, Guilford Press; 1998.
Time Frame: 5 weeks
Population: Children with ADHD who completed the five week diet and parents filled out the ADHD rating scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restricted Diet | Ruse Diet
Number analyzed (Participants) | 15 | 14
units on a scale | 18.0 (10.9) | 21.3 (11.75)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Restricted Diet | Ruse Diet
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 5/15 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restricted Diet (N=15) | Ruse Diet (N=14)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Acid Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Streptococcus Throat Infection (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No